CLINICAL TRIAL: NCT02694588
Title: Systematic Profiling of Anti-inflammatory Drugs for the Detection of Drug- Specific Response Signatures in the Treatment of Chronic Inflammatory Disorders
Brief Title: Clinical and Molecular Phenotyping in IBD
Acronym: Phen_IBD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Mark Ellrichmann, Head of Interdisciplinary Endoscopy, University Hospital Schleswig-Holstein
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Short-Sys-Inflame
Record Dates: First submitted 2015-12-04; First posted 2016-02-29 (Estimated); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: IBD
Keywords: Vedolizumab; Infliximab
MeSH Terms: interventions — Infliximab; vedolizumab

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Infliximab (Active Comparator): 5 mg/kg body weight, week 0/2/6, then every 8 weeks
  Interventions: Drug: Infliximab
- Vedolizumab (Active Comparator): 300 mg, week 0/2/6, then every 8 weeks
  Interventions: Drug: Vedolizumab

INTERVENTIONS:
Drug: Infliximab — HD-endoscopy, CLE, endoscopic ultrasound after application of TNF alpha antibody
  Other Names: Endoscopic assessment after Infliximab
  Arms: Infliximab
Drug: Vedolizumab — HD-endoscopy, CLE, endoscopic ultrasound after application of Anti-Integrin antibody
  Other Names: Endoscopic assessment after Vedolizumab
  Arms: Vedolizumab

SUMMARY:
Inflammatory bowel disease (IBD) and psoriasis (Ps) are common, chronic, immune- mediated barrier diseases with shared inflammatory pathways. Current therapeutic interventions with anti-cytokine antibodies (TNF-α, IL-23/IL-12) reflect the intent to disrupt specific pathways of inflammatory immunopathology. Individual responses to biological treatment can be thereby be exploited in a systems biology approach that employs a targeted mechanism of action (MOA) to decipher molecular signatures of therapeutic responses in the context of a distinct disease entity. Using a translational approach to investigate clinical and molecular phenotypes during therapeutic interference with cytokine signaling and leukocyte trafficking, the investigators aim to trace common and unique signatures of drug- and therapy-specific responses.

Patients will undergo endoscopic evaluation of the mucosal surface and gastrointestinal wall by conventional HD-colonoscopy, endoscopic ultrasound and confocal laser endomicroscopy prior to and during specific therapies with biologicals. In parallel, mucosa samples will be obtained to define molecular phenotypes during the course of therapy.

ELIGIBILITY:
Inclusion Criteria:

* inflammatory bowel disease
* indication for biological therapy

Exclusion Criteria:

* pregnancy, breast feeding
* no written informed consent to participate in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-06; Primary Completion 2018-10 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Mucosal healing week 2 | week 2
  Scoring of mucosal healing according to endoscopic Mayo score at week 2 after initiation of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Schreiber, MD, PhD, Principal Investigator — 00494315971272
Locations (1):
- Medical Department I, University Hospital Schleswig-Holstein, Kiel, Germany

REFERENCES:
- [Derived] Zeissig S, Rosati E, Dowds CM, Aden K, Bethge J, Schulte B, Pan WH, Mishra N, Zuhayra M, Marx M, Paulsen M, Strigli A, Conrad C, Schuldt D, Sinha A, Ebsen H, Kornell SC, Nikolaus S, Arlt A, Kabelitz D, Ellrichmann M, Lutzen U, Rosenstiel PC, Franke A, Schreiber S. Vedolizumab is associated with changes in innate rather than adaptive immunity in patients with inflammatory bowel disease. Gut. 2019 Jan;68(1):25-39. doi: 10.1136/gutjnl-2018-316023. Epub 2018 May 5. PMID 29730603